CLINICAL TRIAL: NCT05905471
Title: Living With a Shoulder Fracture - An Interview Study
Brief Title: Shoulder Fracture Interview Study
Status: Completed | Type: Observational
Sponsor: East Lancashire Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Pauline May, Physiotherapist, East Lancashire Hospitals NHS Trust
Other Study IDs: DEV033
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Proximal Humerus Fracture (Shoulder Fracture)
MeSH Terms: conditions — Shoulder Fractures | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview — Interview study

SUMMARY:
Shoulder fractures are painful injuries and are the third most common fracture in adults. More and more people are having these injuries each year. Problems such as pain, swelling and lack of movement and strength can last for many months and some people never get back to their previous levels of ability with the injured arm. Information that is given to people following this injury can be very difficult to understand. To improve the information that is given to people following a shoulder fracture, it is necessary to understand what it is like to live with a shoulder fracture and what is important to people recovering from this injury.

This study will interview people who have had a shoulder fracture at around one month and around 4-6 months after their injury. These people will be identified from a physiotherapy waiting list. The interviews will explore people's views on their injury, their recovery and how their needs and priorities change over time.

DETAILED DESCRIPTION:
Previous studies have shown that the written information provided to people after a shoulder fracture is varied and complex, and is written by experts without any apparent input from patients. Appropriate information provided at the right time may lead to improved outcomes for patients after a shoulder fracture, which may mean improvements in pain levels and function. Appropriate information may help to increase patients empowerment, which is their ability to use information provided to enable them to make informed decisions regarding their health care and to take a proactive approach in their recovery following an injury such as a shoulder fracture. To ensure that information is accessible and appropriate, it is necessary to understand the experience of living with a shoulder fracture and what is important to those who have sustained this injury.

This study intends to hear the views of people who have had a shoulder fracture both early on (around one month after injury) and later in their recovery (4-6 months after injury). It aims to explore the differing needs and experiences of people at different time points after injury and how their views on recovery change over time.

This may lead to further work on information provision, which may help improve outcomes by providing the right (accessible) information to the right people in the right way at the right time.

ELIGIBILITY:
Inclusion Criteria:

- Aged 18 years or over

Have sustained a proximal humerus fracture and been referred from East Lancashire Hospitals NHS Trust fracture clinic to outpatient physiotherapy

Able and willing to provide written informed consent, as deemed by the Chief Investigator

Exclusion Criteria:

- Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have sustained a shoulder fracture and live in the East Lancashire area.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
To explore how a shoulder fracture impact on daily life | From approximately one to five months post injury
To explore patients' views on recovery at different time points throughout the recovery process. | From approximately one to five months post injury
To explore the needs of patients with respect to information provision following a shoulder fracture. | From approximately one to five months post injury

CONTACTS AND LOCATIONS:
Locations (1):
- East Lancashire Hospitals NHS Trust, Burnley, United Kingdom